CLINICAL TRIAL: NCT00239044
Title: An Open Label Study to Evaluate the Tolerability and Safety of Enteric-coated Mycophenolate Sodium (EC-MPS) in Combination With Cyclosporine Microemulsion (CsA-ME) in Maintenance Renal Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CERL080A2405NL01
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Kidney Transplant Recipients
Keywords: Kidney transplant recipients; Enteric-coated Mycophenolate sodium (EC-MPS)

INTERVENTIONS:
Drug: Enteric-coated Mycophenolate sodium (EC-MPS)

SUMMARY:
To evaluate whether maintenance renal transplant patients on micophenolate mofetil (MMF) can be safely converted to EC-MPS, based on adverse events and acute rejection within 6 months after switching from MMF to a EC-MPS regimen.

ELIGIBILITY:
Inclusion criteria

1. Males and females aged between 18 and 80 years.
2. Recipients of first or secondary cadaveric, living related or unrelated donor kidney transplant at least 6 months after transplantation.
3. Patients currently receiving CsA-ME with MMF , with or without corticosteroids as part of their immunosuppressive regimen for at least 3 months prior to Screening.
4. Patients receiving MMF at reduced dose prior to study entry
5. Patients in a stable condition in terms of graft function (serum creatinine not above 2.3 mg/dL (=204 µmol/L) at screening and at baseline, or not increased by more than 20% at baseline compared to values obtained at screening), no change of immunosuppressive regimen due to graft malfunction, and any known clinically significant physical and/or laboratory changes for at least 2 months prior to enrollment.
6. Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to or at screening. Effective contraception must be used during the trial, and for 6 weeks following discontinuation of the study medication, even where there has been a history of infertility.
7. Patients who are willing and able to participate in the full course of the study and from whom written informed consent has been obtained.

Exclusion Criteria

1. Multi-organ patients (e.g., kidney and pancreas) or previous transplant with any other organ different from kidney (secondary kidney transplant is allowed)
2. Evidence of graft rejection or treatment of acute rejection within two months prior to Screening.
3. Patients with any known hypersensitivity to EC-MPS or other components of the formulation (e.g., lactose)
4. Patients with thrombocytopenia (<75,000/mm3), with an absolute neutrophil count of <1,500/mm3 and/or leukocytopenia (<2,500/mm3), and/or hemoglobin <6.0 g/dL prior to enrollment.
5. Patients who have received an investigational drug within two weeks prior to Screening (i.e., before Day -14 of run-in period).
6. Patients with a history of malignancy within the last five years, except excised squamous or basal cell carcinoma of the skin.
7. Females of childbearing potential who are planning to become pregnant, who are pregnant and/or lactating, who are unwilling to use effective means of contraception
8. Presence of clinically significant infection requiring continued therapy, severe diarrhea, active peptic ulcer disease, or uncontrolled diabetes mellitus that would interfere with the appropriate conduct of the study.
9. Known positive HIV and/or Hepatitis B surface antigen positive.
10. Evidence of drug and/or alcohol abuse.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-12; Primary Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Adverse events and acute rejection within 6 months after switching from MMF to a EC-MPS regimen .

SECONDARY OUTCOMES:
Pharmacokinetic profiles of MMF and EC-MPS.
Patient and graft survival, graft function
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis